CLINICAL TRIAL: NCT01779258
Title: Emollients in the Management of Atopic Dermatitis in Children: Prevention of Flares.
Brief Title: Emollients in the Management of Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V00034 CR 3 13 1B; 2012-004621-24 (EudraCT Number)
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Atopic Dermatitis
Keywords: xerosis; dry skin; dermatitis; eczema; emollient; corticosteroid; flare
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema | interventions — Glycerol; Paraffin; Fluid Therapy; Desonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 2 (Other): Active control arm, Locatop@, Locapred@
  Interventions: Device: Atopiclair®; Drug: Locatop@; Drug: Locapred@
- Group 3 (Other): Absence of emollient treatment, Locatop@, Locapred@
  Interventions: Drug: Locatop@; Drug: Locapred@
- Group 1 (Experimental): glycerol, paraffin (liquid and white soft), Locatop@
  , Locapred@
  Interventions: Drug: glycerol, paraffin (liquid and white soft); Drug: Locatop@; Drug: Locapred@

INTERVENTIONS:
Drug: glycerol, paraffin (liquid and white soft) — 1 application in the morning and in the evening
  Other Names: Dexeryl®
  Arms: Group 1
Device: Atopiclair® — 1 application in the morning, in the afternoon and in the evening
  Arms: Group 2
Drug: Locatop@ — During the Run-In period:
  1 application in the morning and in the evening during a maximum of 21 days
Drug: Locapred@ — During the 3 months study treatment:
  1 application in the evening in case of flare "

SUMMARY:
The purpose of this study is to confirm that emollients play a major role in the maintenance therapy after clearing of inflammatory lesions and can reduce occurrence of flares in children with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 6 years included,
* Presenting with atopic dermatitis, with at least one duly documented flare treated by corticosteroids within the previous 6 months, and presenting a current flare (objective Scoring for Atopic Dermatitis (SCORAD score) is [15-40] at inclusion),
* After treatment of the current flare, patients should have for randomization an Objective SCORAD score < 15, with Xerosis intensity≥ 1 and no subjective signs

Exclusion Criteria:

* Severe form of atopic dermatitis requiring either systemic corticosteroid treatment and/or antibiotic or antiviral treatment and/or hospitalisation,
* Primary bacterial, viral, fungal or parasitic skin infection,
* Ulcerated lesions, acne or rosacea,
* Dermatological disease other than atopic dermatitis which could interfere with the assessment,
* Immunosuppression,

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 347 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one flare over the treatment period | 12 weeks of treatment.
  A flare is defined as following: measurable increased extend or intensity of lesions in less than 2 weeks under continued treatment corresponding to a significant increase in medical score (> 25%) or to the introduction of a new line of therapy(topical corticosteroid).

CONTACTS AND LOCATIONS:
Locations (15):
- Estonia (2):
  - Tallinn
  - Tartu
- France (2):
  - Bordeaux
  - Poitiers
- Vilnius, Lithuania
- Poland (4):
  - Lodz
  - Pruszków
  - Płock
  - Warsaw
- Romania (6):
  - Brasov
  - Bucharest
  - Craiova
  - Iași
  - Sibiu
  - Targu Mureş